CLINICAL TRIAL: NCT05443087
Title: Dosing of Various Multi Kinases Inhibitors Plasma Concentrations for Patients Treated for Their Advanced Digestive Cancer, With the Aim to Determine the Best Optimal Dose for Each Treatment, in the Future
Brief Title: TARGETed Therapy Drug MONITOring in DIGestive Oncology
Acronym: TARGETMONITO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-2104; 2021-A01724-37 (Other: ID-RCB)
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Digestive Cancer; Metastatic Colorectal Cancer; Hepatocellular Carcinoma; GIST; Neuroendocrine Tumors
Keywords: multi kinases inhibitors; therapeutic drug monitoring; pharmacokinetics; pharmacodynamics; advanced digestive cancers
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Carcinoma, Hepatocellular; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Regorafenib - mCRC, GIST, HCC (Experimental): 3 x 30 = 90 patients
  Patients with mCRC, GIST or HCC treated with Regorafenib
  Interventions: Other: Blood sampling to build population pharmacokinetics model
- Everolimus - gepNET (Experimental): 60 patients
  Patients with gepNET treated with Everolimus
  Interventions: Other: Blood sampling to build population pharmacokinetics model
- Sunitinib - pNET, GIST (Experimental): 2 x 30 = 60 patients
  Patients with pNET and GIST, treated with Sunitinib
  Interventions: Other: Blood sampling to build population pharmacokinetics model
- Cabozantinib - HCC (Experimental): 60 patients
  Patients with HCC treated with Cabozantinib
  Interventions: Other: Blood sampling to build population pharmacokinetics model
- Encorafenib - Cetuximab - mCRC (Experimental): 60 patients
  Patients with mCRC treated with the association Encorafenib - Cetuximab
  Interventions: Other: Blood sampling to build population pharmacokinetics model

INTERVENTIONS:
Other: Blood sampling to build population pharmacokinetics model — Determine for each drug plasmatic exposure (Css, trough) through the PopPK model.
  Concentrations measured at the following time points:
  * 1 month after the first treatment administration
  * 2 months after the first treatment administration
  * In case of progression
  * In case of severe toxicities (AESI) related to the drug received

SUMMARY:
Targeted therapy drug monitoring in digestive oncology: Dosage of plasma levels of various multikinase inhibitors (MKI) in patients treated for advanced digestive cancer (gastrointestinal stromal tumor (GIST), metastatic colorectal cancer (mCRC), hepatocellular carcinoma (HCC), gastroenteropancreatic neuroendocrine tumor (gepNET), or pancreatic neuroendocrine tumor (pNET)), with the aim of determine the optimal dose adapted for each patient, in the future.

DETAILED DESCRIPTION:
Phase IV, national, multicenter, open, multi-cohort interventional study:

1. Regorafenib - mCRC, GIST, and HCC = 3x30 = 90 patients
2. Everolimus - gepNET = 60 patients
3. Sunitinib - pNET and GIST = 60 patients
4. Cabozantinib - HCC = 60 patients
5. Encorafenib-cetuximab - mCRC = 60 patients

The patients included will be treated and followed according to standard practice (national recommendations and according to the summary of product characteristics (SmPC) of each molecule). According to the cohort, a maximum of 1 to 2 blood tubes will be taken at different times during the study: at baseline, then 1 month after the start of treatment, then 2 months after the start of treatment, if an adverse event of specific interest (AESI) occurs, and in case of progressive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years or over
2. Advanced digestive cancer (histologically confirmed or confirmed by imaging for HCC) for which a standard treatment (according to each drug SmPC and as per standard of care) planned with:

   * Regorafenib for GIST, mCRC, and HCC,
   * Everolimus for gepNET,
   * Sunitinib for pNET or GIST,
   * Cabozantinib for HCC,
   * Encorafenib - cetuximab for mCRC
3. Life expectancy of greater than 3 months - at the discretion of the investigator
4. Measurable disease according to tumor evaluation criteria as per local practice (Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, etc.)
5. Patients must be affiliated to a Social Security System (or equivalent)
6. Patient must have signed a written informed consent form prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.

Exclusion Criteria:

1. Other concomitant anticancer systemic treatment (chronic chemotherapy, antitumor hormone therapy or immunotherapy) than the one studied
2. Unresolved toxicity higher than NCI-CTCAE v5.0 Grade 1 attributed to any prior therapy/procedure excluding alopecia and peripheral neuropathy
3. Prior treatment with the same MKI molecule(s) planned to be given in the cohort. If different MKI molecules (from the one(s) planned in the study) have been previously taken, a wash out period of 2 weeks before treatment should be observed.
4. Other invasive malignancies either currently active or active in the last 3 years, except adequately treated in situ carcinoma of the cervix and basal or squamous cell carcinoma of the skin
5. Any condition that may jeopardize patient participation in the study as well as non contraception for male and female with child-bearing potential, pregnancy or breast feeding.
6. Patient unwilling or unable to comply with the medical follow-up required by the standard treatment taken (including PK sampling during treatment phase and vital status collection during follow-up phase) because of psychosocial, familial, social or geographical reasons
7. Participation in another clinical study with an investigational medicinal product during the last 30 days prior to inclusion and during the present study (except if patient is included in the control arm, with placebo or with a product which have a marketed authorisation, used as per the SmPC for the given indication)
8. Patient deprived of their liberty or under protective custody or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Trough concentration (Ctrough) | From inclusion untill the end of treatment up to 4 years
  Trough concentration (Ctrough) shows the blood concentration reached by a drug immediately before the next dose is administered, once steady state has been attained. It can also be defined as the minimal drug concentration in the patient's body. Plasmatic measures will be performed by liquid chromatography with tandem mass spectrometry after protein precipitation by acetonitrile.

SECONDARY OUTCOMES:
Progression-free survival | 4 years
  Progression-free survival (PFS) is the lenght of the time between inclusion and the first event of disease progression or death whatever the cause.
Overall survival | 4 years
  Overall survival (OS) is the lenght of time between inclusion and death whatever the cause.
Objective response rate | 4 years
  Objective response rate (ORR) is the percentage of patients with a best response during treatment being either complete response (CR) or partial response (PR).
Disease control rate | 4 years
  Disease control rate (DCR) is defined as the percentage of patients with a best response during treatment being either CR, PR, or Stable Disease (SD).
Safety: drug toxicity | Throughout study completion, up to 4 years
  Drug toxicity occurrence related to standard treatment will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0. NCI-CTCAE is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
  Only AE of Specific Interest (AESI) will be collected.
  An AESI is an AE related to treatment that is:
  * G3 or G4 according to NCI-CTCAE version 5.0, or
  * Leading to treatment modification (dose reduction or treatment interruption), or
  * Categorized as serious adverse event (SAE) by the investigator, or
  * Considered as clinically significant by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: David MALKA, Dr, Principal Investigator — Gustave ROUSSY - VILLEJUIF
Locations (29):
- France (29):
  - CHU d'Amiens Pcardie - Hopital Sud, Amiens
  - CH d'Auxerre, Auxerre
  - Institut du Cancer Avignon - Institut Sainte Catherine, Avignon
  - CH de Bayeux - Onconormandie, Bayeux
  - Centre Jean Perrin, Clermont-Ferrand
  - Hôpital Beaujon APHP, Clichy
  - Centre Georges Francois Leclerc, Dijon
  - Institut de Cancérologie de Bourgogne, Dijon
  - CH Eure Seine - Hopital d'Evreux Vernon, Évreux
  - Centre Oscar Lambret, Lille
  - Groupement des hôpitaux de l'Institut Catholique de Lille - Hôpital Saint Vincent de Paul, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Européen Marseille, Marseille
  - CHRU de Nancy - Hôpital de Brabois Adulte, Nancy
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - APHP Pitié Salpétrière, Paris
  - Hôpital Saint Joseph, Paris
  - Institut Mutualiste de Montsouris, Paris
  - Hôpital Privé des Côtes d'Armor - SAS, Plérin
  - CHU de Poitiers, Poitiers
  - CHU de Reims - Hôpital Robert Debré, Reims
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - CHU Rouen - Hôpital Charles Nicolle, Rouen
  - CH Saint Malo - Hôpital Broussais, St-Malo
  - ICANS, Strasbourg
  - CHU de Tours, Tours
  - Gustave Roussy, Villejuif